CLINICAL TRIAL: NCT03219125
Title: Bone Marrow Adiposity and Fragility Fractures in Postmenopausal Women: a Case-control Study
Brief Title: Bone Marrow Adiposity and Fragility Fractures in Postmenopausal Women
Acronym: ADIMOS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_44; 2017-A00472-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2020-11

CONDITIONS: Fractures, Bone; Bone Marrow Disease; Fat Disorder; Adiposity
Keywords: marrow adipose tissue; bone marrow adiposity
MeSH Terms: conditions — Fractures, Bone; Bone Marrow Diseases; Lipid Metabolism Disorders; Obesity | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (cases): occurence of incident major osteoporotic fracture less than 12 weeks
  Interventions: Device: Dixon Magnetic Resonance Imaging
- Group 2 (controls): no history of fragility fracture
  Interventions: Device: dual-energy X-ray absorptiometry (DXA)

INTERVENTIONS:
Device: Dixon Magnetic Resonance Imaging — MRI of the lumbar spine (L1 to L4) and hip (non-dominant) for the measurement of Ad Med. (In%) by the DIXON sequence.
  Groups: Group 1 (cases)
Device: dual-energy X-ray absorptiometry (DXA) — Subjects will undergo DXA scan to assess total body (less head) and lumbar spine bone mineral density.
  Groups: Group 2 (controls)

SUMMARY:
The purpose is to determine in a case-control study if an association exist between bone marrow adiposity and fragility fractures in post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women : 50-90 years old
* Group 1 (cases) : occurence of incident major osteoporotic fracture less than 12 months
* Group 2 (controls) : no history of fragility fracture

Exclusion Criteria:

* Implants that are contraindicated for the magnetic resonance (MR) examination.
* Implants that might create a health risk or other problem during an MR exam include: 1) cardiac pacemaker or implantable defibrillator, 2) catheter that has metal components that may pose a risk of a burn injury, 3) a ferromagnetic metal clip placed to prevent bleeding from an intracranial aneurysm, 4) an implanted medication pump (such as that used to deliver insulin or a pain-relieving drug), and 5) a cochlear implant.
* body mass index [BMI] >38 kg/m2, weight >140 kg
* Disease or current use of medications known to affect bone density, including oral glucocorticoids, treatments for osteoporosis (bisphosphonates, raloxifene, calcitonin, or PTH), hormone therapy.
* Chronic kidney disease with DFG <30 ml/mn

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-menopausal women
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Bone marrow fat content at lumbar spine | 24 months
  Total bone marrow fat content (percentage) at lumbar spine (L1-L4) measured with magnetic resonance imaging

SECONDARY OUTCOMES:
Bone marrow fat content at total hip | 24 months
  Total bone marrow fat content (percentage) at total hip measured with magnetic resonance imaging
Bone mineral density at lumbar spine | 24 months
  Bone mineral density (g/cm2) at lumbar spine (L1-L4) measured by DXA
Bone mineral density at total hip | 24 months
  Bone mineral density (g/cm2) at total hip measured by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Julien Paccou, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No